CLINICAL TRIAL: NCT03704233
Title: The Diagnostic Yield and Safety of Transbronchial Cryobiopsy in Diffuse Parenchymal Lung Diseases: a Prospective, Multicenter, Real World Study
Brief Title: The Diagnostic Yield and Safety of Transbronchial Cryobiopsy in Diffuse Parenchymal Lung Diseases
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Guangzhou Institute of Respiratory Disease (Other)
Responsible Party: Principal Investigator, ShiYue Li, Director of Department of Respiratory Medicine, Guangzhou Institute of Respiratory Disease
Other Study IDs: 2018-03-13
Record Dates: First submitted 2018-09-25; First posted 2018-10-12 (Actual); Last update posted 2019-03-07 (Actual); Status verified 2019-03

CONDITIONS: Diffuse Parenchymal Lung Diseases
Keywords: Transbrochial cryobiopsy; Diffuse parenchymal lung diseases; Diagnosis
MeSH Terms: conditions — Lung Diseases, Interstitial; Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cryobiopsy: Transbronchial cryobiopsy is performed in patients with undefined diffuse parenchymal lung diseases, and assess the diagnostic yield and safety.
  Interventions: Procedure: Transbronchial cryobiopsy

INTERVENTIONS:
Procedure: Transbronchial cryobiopsy — Transbronchial cryobiopsy procedure

SUMMARY:
The Diagnostic yield and Safety of transbronchial cryobiopsy in the diagnosis of diffuse parenchymal lung diseases are investigated in this multicenter, prospective and real world study.

ELIGIBILITY:
Inclusion Criteria:

1. The patients are admitted in the institution as DPLD, while undefined after thorough history collection, laboratory examination and radiological data.
2. Transbronchial cryobiopsy(TBCB) is indicated by clinicians for definitive diagnosis and patients are content with the examination with agreement signed.
3. Blood gas analysis, routine blood test, ECG examination, coagulation function, immunological examination, chest HRCT, and liver/kidney function test have been completed.

Exclusion Criteria:

1. The radiological data indicates non-DPLD
2. The clinical examinations mentioned above are not completed.
3. The patient cannot endure or does not agree the procedure.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Inpatients
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2020-10-20 (Estimated); Study Completion 2021-10-20 (Estimated)

PRIMARY OUTCOMES:
Diagnotic yield | two weeks
  Percentage of definitive pathological diagnosis by transbronchial cryobiopsy, the alteration of original diagnosis after transbronchial cryobiopsy

SECONDARY OUTCOMES:
Complication rate | 12 weeks
  Incidence of bleeding, pneumothorax (during the procedure and within 7 days after the intervention) and exacerbations of DPLD related to the transbronchial cryobiopsy (in 12 weeks).

CONTACTS AND LOCATIONS:
Overall Officials: Shiyue Li, Study Chair — Guangzhou Institute of Respiratory Disease, The First Affiliated Hospital of Guangzhou Medical University
Locations (26):
- China (26):
  - AnHui Chest Hospital, Hefei, Anhui
  - China-Japan Friendship Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Xiamen Second Hospital, Xiamen, Fujian
  - Guangdong General Hospital, Guangzhou, Guangdong
  - the First Affiliated Hospital Sun Yat-sen University, Guangzhou, Guangdong
  - Guangzhou Institute of Respiratory Disease, The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Southern Medical University Nanfang Hospital, Guangzhou, Guangdong
  - Peking University Shenzhen Hospital, Shenzhen, Guangdong
  - Shenzhen Guangming New District People's Hospital, Shenzhen, Guangdong
  - Affiliated Zhongshan Hospital of Guangdong Medical University, Zhongshan, Guangdong
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - The Central Hospital Of WuHan, Wuhan, Hubei
  - Department of Respiratory and Critical Care Medicine，Tongji Hospital，Tongji Medical College，Huazhong University of Science and Technology, Wuhan, Hubei
  - People's Hospital of Hunan Province, Changsha, Hunan
  - XiangYa Hospital Central South University, Changsha, Hunan
  - Dalian Muncipal Central Hospital Affiliated of Dalian Medical University, Dalian, Liaoning
  - The First Hospital of China Medical University, Shengyang, Liaoning
  - Shanghai Chest Hospital, Shanghai, Shanghai Municipality
  - Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality
  - Renji Hospital Affiliated to Shanghai Jiao Tong University, Shanghai, Shanghai Municipality
  - Xi'an chest hospital, Xi’an, Shanxi
  - West China School of Medicine/West China Hospital of Sichuan University, Chengdu, Sichuan
  - MianYang Central Hospital, Mianyang, Sichuan
  - China Medical University Hospital, Taizhong, Taiwan
  - The first Hospital of Jiaxing, Jiaxing, Zhejiang

REFERENCES:
- [Derived] Chen X, Li J, Luo F, Tao F, Zhang X, Wu Y, Xu P, Ke M, Long F, Liu L, Lv L, Liao H, Gu Y, Liu Z, Tan X, Guo S, Hu Y, Yang H, Zhou Y, Zhou H, Ye Y, Chen D, Li S. The application of transbronchial cryobiopsy in interstitial lung disease: a prospective, multicenter, real-world study. Ann Transl Med. 2021 Nov;9(22):1645. doi: 10.21037/atm-21-3461. PMID 34988154